CLINICAL TRIAL: NCT02813395
Title: Immediate Effects of Low-level Laser Therapy (808nm) on Neuromuscular Performance After Muscle Fatigue: Randomized-blinded Clinical Trial
Brief Title: Laser Therapy on Neuromuscular Performance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal do Rio Grande do Norte (Other)
Responsible Party: Principal Investigator, Jamilson Simões Brasileiro, PhD, Universidade Federal do Rio Grande do Norte
Allocation: Randomized | Model: Parallel | Masking: Triple
Other Study IDs: RMV2016
Record Dates: First submitted 2016-06-21; First posted 2016-06-27 (Estimated); Last update posted 2016-06-27 (Estimated); Status verified 2016-06

CONDITIONS: Fatigue
MeSH Terms: conditions — Fatigue | interventions — Low-Level Light Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (4):
- Control group (No Intervention): Volunteers remained at rest before and after the fatigue protocol.
- Placebo group (Placebo Comparator): Volunteers were subjected to laser application simulation for approximately four minutes with a second pen of the laser device, which was disconnected and did not effectively irradiate energy.
  Interventions: Device: Placebo Laser
- Laser before (Experimental): Volunteers received effective application of laser before fatigue protocol.
  Interventions: Device: Low Level Laser Therapy
- Laser after (Experimental): Volunteers received effective application of laser after fatigue protocol.
  Interventions: Device: Low Level Laser Therapy

INTERVENTIONS:
Device: Low Level Laser Therapy — Low Level Laser Therapy was applied at four points to the dominant upper limb of the volunteers on the muscle belly of the biceps. Delineation was done using a measuring tape from the elbow joint line to the acromion marked at points corresponding to 20%, 30%, 40% and 50% of this distance, focusing the application on the muscle belly region, thereby excluding the tendinous region.
  An 808 nm equipment was used for applying laser therapy, with a power of 100 mW and total energy of 20 J.
  Arms: Laser after; Laser before
Device: Placebo Laser — Laser application simulation with a second pen of the laser device, which was disconnected and did not effectively irradiate energy.
  Arms: Placebo group

SUMMARY:
Objective: Investigating the immediate effects of Low Level Laser Therapy (LLLT) on neuromuscular performance in healthy subjects after an induced muscle fatigue protocol. Methods: Eighty volunteers of both genders aged between 18 and 28 years underwent a preliminary evaluation using surface electromyography and isokinetic dynamometer of the flexor muscles of the elbow. The subjects were randomly allocated into 4 groups: G1 was control group; G2 placebo; G3 laser applied before fatigue protocol; and G4 immediately after. Muscular fatigue protocol consisted of 30 maximal concentric isokinetic contractions at 120°/s of the elbow flexor muscles. An 808 nm equipment was used for applying laser therapy, with a power of 100 mW and total energy of 20 J. Volunteers were reassessed after interventions.

ELIGIBILITY:
Inclusion Criteria:

* Being between 18-28 years of age, having no pain in the shoulder area, elbow or hand, and not having suffered any to injury to the assessed upper limb in the last six months.

Exclusion Criteria:

* Presenting pain that prevented the completion of the evaluation, subjects whose data were improperly recorded or if the volunteer withdrew from the study.

Ages: 18 Years to 28 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2014-04; Primary Completion 2015-03 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Peak torque normalized by body weight | Change from baseline to one hour.

CONTACTS AND LOCATIONS:
Locations (1):
- Federal University of Rio Grande do Norte, Natal, Rio Grande do Norte, Brazil